CLINICAL TRIAL: NCT06960707
Title: Prospective Randomized Trial of Two Versus One Week Accelerated Radiotherapy (PRATO)
Brief Title: Two Versus One Week Breast Radiotherapy (RT)
Acronym: PRATO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-01028391
Record Dates: First submitted 2025-04-28; First posted 2025-05-07 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: Accelerated Radiotherapy; Prone Position; Adjuvant Setting; Non-Inferiority; Concomitant Boost
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ARM 1-2600 cGy in 5 fractions whole breast radiotherapy (Experimental): Patients randomized to ARM 1 will receive 2600 cGy in 5 fractions whole breast radiotherapy over one week
  Interventions: Radiation: Radiation therapy - 1 week
- ARM 2- 3200 cGy in 10 fractions with a concomitant tumor bed boost to 3600 cGy (Experimental): Patients randomized to ARM 2 will receive 3200 cGy in 10 fractions with a concomitant tumor bed boost to 3600 cGy.
  Interventions: Radiation: Radiation therapy - 2 weeks

INTERVENTIONS:
Radiation: Radiation therapy - 1 week — 2600 cGy whole breast radiotherapy in five fractions (Arm 1) over 1 week
  Arms: ARM 1-2600 cGy in 5 fractions whole breast radiotherapy
Radiation: Radiation therapy - 2 weeks — 3200 cGy whole breast radiotherapy with a concomitant tumor bed boost to 3600 cGy in 10 fractions (Arm 2) over 2 weeks. In Arm 2, if no cavity is visible due to oncoplastic surgery, we will deliver 32 Gy to the whole breast only, without a boost.
  Arms: ARM 2- 3200 cGy in 10 fractions with a concomitant tumor bed boost to 3600 cGy

SUMMARY:
This study is comparing two different radiation therapy approaches for early breast cancer to see which one is better for patients. One group will receive radiation over one week (based on the FAST-FORWARD trial), and the other group will receive radiation over two weeks with an extra focused dose (called a "concomitant boost"). The study will look at how the treatments affect side effects, breast appearance, and cancer control in the breast. It also aims to find out if the two-week treatment does a better job at preventing cancer from coming back in the breast over the long term.

DETAILED DESCRIPTION:
Radiotherapy: one week (Arm 1) 2600 cGy in 5 fractions whole breast radiotherapy over one week versus 2 weeks (Arm 2), 3200 cGy in 10 fractions with a concomitant tumor bed boost to 3600 cGy. In Arm 2, if no cavity is visible due to oncoplastic surgery, we will deliver 32 Gy to the whole breast only, without a boost.

Hypothesis: A regimen of whole breast radiotherapy to 2600 in five fractions, the current UK standard for early breast cancer (Arm 2), is not inferior to 3200cGy with a concomitant tumor bed boost to 3600 cGy in 10 fractions (Arm 1), in terms of acute toxicity and long-term fibrosis, breast cosmesis and local control at 2 and 5 years. It will also test the hypothesis of superior local control at 10 years in Arm 2 compared to Arm 1.

ELIGIBILITY:
Inclusion Criteria:

1. Women status post segmental mastectomy.
2. If unilateral, pT1-2 breast cancer excised with negative margins.
3. If bilateral, pT1-2 breast cancer excised with negative margins AND/OR pTis excised with negative margins.
4. Clinically N0 (cN0 as determined by ultrasound/SOUND criteria) or pN0-1 or Nx or sentinel node negative.
5. Ductal carcinoma in situ DCIS with negative margins (no DCIS on inked margins).
6. Women with previous contralateral treated breast cancer can be enrolled in the trial.

Exclusion Criteria:

1. Previous radiation therapy to the ipsilateral breast.
2. >90 days from last surgery, unless s/p adjuvant chemotherapy.
3. >60 days from last chemotherapy.
4. Male breast cancer.
5. Ongoing treatment for severe autoimmune disease.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 400 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of RT-related acute toxicity | 1 month
  The rate of RT-related acute toxicity is defined as cumulative acute toxicity events from the start of radiation treatment to 1 month follow up post RT. The toxicities will be graded by the research nurses assigned to the study according to Common Terminology Criteria for Adverse Events, version 5.0.

SECONDARY OUTCOMES:
The long-term evaluations at 2 years of fibrosis based on LENT/SOMA | 24 months
  The number of subjects scoring Grades 1 through 4 using the LENT/SOMA (Late Effects Normal Tissues (LENT)-Subjective, Objective, Management, Analytic (SOMA)) system will be reported.
  The patients will grade the following items based on the following scale:
  1. Mild
  2. Moderate
  3. Severe
  4. Life-threatening
The long-term evaluations at 2 years of breast cosmesis | 24 months
  Patient self-reported breast cosmesis will be assessed using the BCTOS questionnaire (Breast Cancer Treatment Outcome Scale).The number of subjects scoring Grades 1 through 4 will be reported. The patients will grade the following items based on the following scale:
  1. = No difference between treated and untreated breast/area
  2. = Slight difference
  3. = Moderate difference
  4. = Large difference
The long-term evaluations at 2 years of local control | 24 months
  Number of subjects with Local control at 2 years will be extracted from the medical record, and can be derived from clinical reports from medical, surgical or radiation oncologists as well as from the primary care doctor who is following the patient.
The long-term evaluations at 5 years OF fibrosis based on LENT/SOMA | 60 months
  The number of subjects scoring Grades 1 through 4 using the LENT/SOMA (Late Effects Normal Tissues (LENT)-Subjective, Objective, Management, Analytic (SOMA)) system will be reported.
  The patients will grade the following items based on the following scale:
  1. Mild
  2. Moderate
  3. Severe
  4. Life-threatening
The long-term evaluations at 5 years of breast cosmesis | 60 months
  Patient self-reported breast cosmesis will be assessed using the BCTOS questionnaire (Breast Cancer Treatment Outcome Scale). The number of subjects scoring Grades 1 through 4 will be reported. The patients will grade the following items based on the following scale:
  1. = No difference between treated and untreated breast/area
  2. = Slight difference
  3. = Moderate difference
  4. = Large difference
The long-term evaluations at 5 years of local control. | 60 months
  Number of subjects with Local control at 5 years will be extracted from the medical record, and can be derived from clinical reports from medical, surgical or radiation oncologists as well as from the primary care doctor who is following the patient.
Superior local control at 10 years | 120 months
  Number of subjects with Local control at 10 years will be extracted from the medical record, and can be derived from clinical reports from medical, surgical or radiation oncologists as well as from the primary care doctor who is following the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia C. Formenti, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- United States (3):
  - Brooklyn Methodist Hospital, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - New York-Presbyterian Weill Cornell Medical College, New York, New York

IPD SHARING:
Plan to Share IPD: No